CLINICAL TRIAL: NCT03480854
Title: Improving Quality and Value of Multiple Sclerosis Care at the Microsystem Level: The Multiple Sclerosis Continuous Quality Improvement (MSCQI) Collaborative
Brief Title: The Multiple Sclerosis Continuous Quality Improvement (MSCQI) Collaborative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: MGH Multiple Sclerosis Clinic (Unknown); University of Vermont (Other); Neurology Associates Multiple Sclerosis Center of Greater Orlando (Unknown); Concord Hospital (Other)
Responsible Party: Principal Investigator, Brant J. Oliver, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D16181; US-MSG-15-10917 (Other Grant/Funding Number: Biogen)
Record Dates: First submitted 2017-05-18; First posted 2018-03-29 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Quality Improvement

STUDY DESIGN:
Intervention Model Description: This is a two-part prospective study to be conducted over 3 years with option to extend to 5 years. In Year 1, we will gather baseline performance data from participating MS clinics (microsystems), create a combined MSCQI systems-level database, and conduct analyses of performance variation and benchmarking. In the second part of the study (Years 2-3), we will investigate the effect of Continuous Quality Improvement interventions on primary endpoints and selected secondary measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Analysis (No Intervention): To conduct studies of variation in performance across microsystems and to utilize benchmarking analyses to identify top performers.
- The effect of continuous quality improvements (CQI) (Experimental): To study the comparative improvement of selected primary process performance indicators (DMT and MRI process measures) over a 3 year period (Years 2-3) in microsystems receiving CQI interventions versus those not receiving CQI intervention, and between two different CQI intervention types (IHI Breakthrough Series and Patient Centered Medical Home).
  Interventions: Other: Quality Improvement

INTERVENTIONS:
Other: Quality Improvement — Randomly selected sites will receive one of two system level improvement approaches; 1) patient centered specialty medical home certification 2) IHI Breakthrough Series improvement approach with professional improvement coaching.
  Arms: The effect of continuous quality improvements (CQI)

SUMMARY:
To establish the first systems level continuous quality improvement (CQI) collaborative for multiple sclerosis (MS) in the United States, to conduct benchmarking analyses and assessments of geographic variation in MS care quality and value, and study the effect of CQI interventions on improvement of selected performance (quality) indicators.

DETAILED DESCRIPTION:
This is a three year study which employed a step-wedge randomized design which exposed three of four participating centers to a healthcare QI intervention during the 3 year period. Each of the centers exposed to an intervention served as its own control during a baseline pre-intervention period during the first year of the study. The fourth site served as a longitudinal control for comparison to the other three centers exposed to a QI intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older with documented clinically confirmed MS who are followed by one of the participating MS centers.

Exclusion Criteria:

* Candidates will be excluded from study entry if they are unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Disease modifying therapy utilization | every 12 weeks for a period of 36 months
  The percentage of eligible MS patients on disease modifying therapy (DMT access), which is operationally defined as the total number of eligible patients on DMT/the total number of patients seen per quarter at a participating center for whom DMT is an appropriate treatment option.

SECONDARY OUTCOMES:
Clinical outcome for Depression | every 12 weeks for a period of 36 months
  patient reported outcome of The Effects of Your MS (PHQ-9)
Clinic Outcome for Anxiety | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Anxiety survey
Clinic Outcomes on Cognitive Function | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Cognitive Function survey
Clinic Outcomes on mobility | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Lower Extremity Function (Mobility) survey
Clinic Outcomes on fine motor skills and activities of daily living | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Upper Extremity Function (Fine Motor, ADL) survey
Clinic Outcomes on stigma associated with MS | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Stigma survey
Clinic Outcomes on ability to participate in social roles and activities | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Ability to Participate in Social Roles and Activities survey
Clinic Outcomes on satisfaction with social roles and activities | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Satisfaction with Social Roles and Activities survey
Clinic Outcomes for sleep disturbance | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Sleep Disturbance survey
Clinic Outcomes for communication | every 12 weeks for a period of 36 months
  patient reported outcome of Neuro-QOL: Communication survey
Clinic Outcomes for Vitamin D levels in MS patients | every 12 weeks for a period of 36 months
  patient reported outcome of Vitamin D Level survey
Clinic Outcomes for fatigue | every 12 weeks for a period of 36 months
  patient reported outcome of PROMIS Fatigue MS survey
Clinic Outcomes for assesment of patient health status | every 12 weeks for a period of 36 months
  patient reported outcome of Brief Appraisal Inventory survey
Clinic Outcomes for satisfaction of treatment by medication | every 12 weeks for a period of 36 months
  patient reported outcome of Treatment Satisfaction Questionnaire for Medication (TSQM-9) survey
Clinic Outcomes for the effects of MS on the patient | every 12 weeks for a period of 36 months
  patient reported outcome of The Effects of Your MS (PDDS) survey
Clinic Outcomes for the presence of a MS relapse | every 12 weeks for a period of 36 months
  patient reported outcome of My MS Relapse Evaluation survey
Clinic Outcomes reporting of MS patient daily symptoms | every 12 weeks for a period of 36 months
  patient reported outcome of the Daily Symptoms survey
Medical History | every 12 weeks for a period of 36 months
  data regarding medical history reported by the patient
Hospitalization | every 12 weeks for a period of 36 months
  data regarding hospitalization reported by the patient
Demographic information | every 12 weeks for a period of 36 months
  data regarding demographics reported by the patient
Medication | every 12 weeks for a period of 36 months
  survey data regarding medication use reported by the patient
MRI utilization | every 12 weeks for a period of 36 months
  survey data regarding number of MRIs reported by the patient
Exercise | collected daily and summarized annually.
  survey data regarding daily exercise
System level measure the patient experience for ambulatory care. | every 12 weeks for a period of 36 months
  Health care quality assessment collected through the Aggregated Clinician and Group Survey to assess patient experience in ambulatory care.
System level measure of Health Care Quality | every 12 weeks for a period of 36 months
  Patient determined disease steps survey

CONTACTS AND LOCATIONS:
Overall Officials: Brant J Oliver, PhD, Principal Investigator — Dartmouth Hitchock
Locations (4):
- United States (4):
  - Neurology Associates of Greater Orlando, Maitland, Florida
  - Massachusetts General Hospital Multiple Sclerosis Center, Boston, Massachusetts
  - Concord Hospital, Concord, New Hampshire
  - University of Vermont Multiple Sclerosis Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No